CLINICAL TRIAL: NCT01058980
Title: ADenosine Following Pulmonary Vein Isolation to Target Dormant Conduction Elimination: the ADVICE Trial
Acronym: ADVICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Abbott Medical Devices (Industry); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Laurent Macle, Chair, ADVICE Study, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICM 08-1067
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Paroxysmal Atrial Fibrillation; Pulmonary Vein Isolation; Dormant Pulmonary Vein Conduction
Keywords: catheter ablation; atrial fibrillation; adenosine
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dormant PV conduction (Active Comparator): After PVI, dormant conduction will be evaluated using intravenous adenosine. If dormant conduction is present, the patients will be randomized to two parallel groups:
  * Group 1: No additional ablation
  * Group 2: Additional ablation until elimination of dormant conduction.
  Interventions: Procedure: Additional ablation until elimination of dormant conduction; Procedure: No additional ablation
- No dormant PV conduction (Active Comparator): If no dormant conduction is documented, patients will be selected in a random fashion to be included in a registry (follow-up as planned for group 1 and 2 above). The registry group will allow for further assessment of the role of dormant conduction as a predictor of AF recurrence by comparing the success rate after ablation in patients without dormant conduction with those of Group 1 and 2.
  Interventions: Procedure: Registry group; Procedure: Usual medical care

INTERVENTIONS:
Procedure: Additional ablation until elimination of dormant conduction — Additional RF energy will be delivered at sites of re-conduction on the circular mapping catheter in each PV. Abolition of the dormant conduction will then be assessed by repeated injections of adenosine using the same doses previously used to reveal dormant conduction. Additional ablation as described will be performed until re-injection of adenosine shows no re-conduction in any of the PV.
  Arms: Dormant PV conduction
Procedure: No additional ablation — Presence of dormant PV conduction, no additional ablation.
  Arms: Dormant PV conduction
Procedure: Registry group — Among those who will be found not to have the presence of dormant conduction, and within each site, three-quarters of the patients will be randomly selected to be included in the registry group.
  Arms: No dormant PV conduction
Procedure: Usual medical care — Clinical follow-up will be performed according to the regular follow-up after AF ablation procedures in each of the participating centers. No data will be collected after discharge.One-fourth of the patients will be randomly selected to be included in the usual medical care group.
  Arms: No dormant PV conduction

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder, impairs quality of life and increases stroke risk and mortality. Despite advances in medical treatment, AF remains uncontrolled in many patients. In many patients, AF is initiated by abnormal electrical impulses from the pulmonary veins. A catheter ablation procedure called pulmonary vein isolation (PVI) has therefore been developed, using heat to isolate the PV foci from the heart. PVI is very effective, but must be repeated in up to 50% of cases because the foci isolation is not permanent after initial PVI. The intravenous administration of a drug called adenosine during the PVI procedure can unmask residual conduction that would otherwise remain unnoticed, so-called "dormant conduction". In our experience, additional ablation guided by adenosine reduces AF recurrence and the need for a repeat PVI procedure. However, the adenosine-guided approach has not yet been proven as standard therapy. The present study, to be conducted at 15 clinical centres in Canada, Europe and Australia is therefore intended to evaluate the efficacy of adenosine-guided ablation to prevent AF recurrence. Five hundred twenty-six patients will be included in the study, which should be completed within 2 years. In all patients, the presence of dormant conduction will be tested with adenosine during PVI. If dormant conduction is observed, additional ablation will be performed in half of these patients selected randomly. If there is no dormant conduction, randomly selected patients will be followed in a registry. If the adenosine-guided approach is demonstrated to improve the success rate of PVI procedures, it should become the standard approach for a "permanent cure" of AF, and therefore benefit patients by reducing arrhythmia recurrence, hospitalizations and the need for repeat interventions.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), the most frequently treated cardiac arrhythmia, impairs quality of life and increases stroke risk and mortality. Despite advances in antiarrhythmic drug therapy, AF remains uncontrolled in many patients. More effective measures to prevent, treat and potentially cure AF are needed. Ectopic foci originating from pulmonary veins (PVs) initiate AF in many patients. PV isolation (PVI), in which PV conduction is eliminated by catheter ablation, has emerged as an effective treatment in selected patients. However AF recurs in up to 50%, due to recovery of PV conduction. Dormant PV conduction (PV conduction suppressed at time of PVI with subsequent recovery) has been proposed to explain recurrences. We demonstrated that adenosine can restore conduction in viable PVs after attempted PVI by activating outward K+-currents, leading to selective hyperpolarization of PV cardiomyocytes and removal of voltage-dependent Na+-channel inactivation. Thus, adenosine can be used to differentiate permanent PV-atrial block from dormant PV conduction and to identify the need for additional ablation. We recently performed a pilot study in 47 patients, in whom adenosine was used to guide additional ablation. Results were compared to 47 historical controls. Dormant conduction was observed in 55% of patients undergoing PVI and additional adenosine-guided ablation decreased the AF recurrence rate from 49% to 21%. An adequately-powered prospective randomized controlled clinical trial is required to confirm these findings.

The primary objective of the proposed ADVICE trial is to evaluate the impact of adenosine-guided PVI in preventing AF recurrences among patients with paroxysmal AF. We hypothesize that a PVI ablation strategy that incorporates elimination of dormant conduction unmasked by intravenous adenosine will decrease symptomatic AF recurrence compared to standard PVI, without incurring significant additional risk. This prospective randomized study will be conducted at 15 clinical centers in Canada, Europe and Australia. Patients with paroxysmal AF referred for PVI will be recruited. Standard PVI will be performed in all patients until elimination of PV conduction. All patients will subsequently receive intravenous adenosine in an attempt to unmask dormant conduction. If dormant conduction is elicited, patients will be randomized to no further ablation (Group 1; control) or additional adenosine-guided ablation until dormant conduction is abolished (Group 2; adenosine-guided PVI). If no dormant conduction is revealed, randomly selected patients will be followed in a registry to further assess the role of dormant conduction as a predictor of AF recurrence. Portable electrocardiographic monitors will be provided to all patients. The primary outcome will be the time to first documented symptomatic AF episode post-PVI based on an intention-to-treat analysis. Since symptomatic AF recurrence is anticipated in 45% of controls, 210 patients with dormant conduction are required in order to be able to detect a difference of 20%, with a power of at least 85%. Assuming the presence of dormant conduction in a minimum of 40% of patients after standard PVI, 526 patients will be enrolled in the study. Enrolment is expected to be completed within 12 months, with all patients followed for 12 months.

Demonstrated superiority of an adenosine-guided PVI ablation strategy would represent a major advancement in refining the interventional approach for AF. The ADVICE trial carries the potential, therefore, to alter the standard of care and benefit patients with AF by reducing arrhythmia recurrence, hospitalizations and the need for repeat interventions

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Paroxysmal AF for at least 6 months with at least 3 symptomatic episodes (using patient history) during the previous 6 months
* Patients must be felt to be candidates for AF ablation based on AF that is symptomatic and refractory or intolerant to at least one class 1 or 3 antiarrhythmic agent.
* Documentation of at least one episode of AF on 12 lead ECG, TTM or Holter monitor within 12 months of randomization in the trial
* Patients must be on continuous anticoagulation with warfarin (INR 2-3) or fractionated subcutaneous heparin for >4 weeks prior to the ablation or they have undergone a recent (less than 48 hours before planned ablation) transoesophageal echocardiogram to exclude left atrial thrombus.
* Patients must provide written informed consent to participate in the clinical trial.

Exclusion Criteria:

* Contraindications to oral anticoagulants
* History of any previous ablation or surgical maze for AF
* Intracardiac thrombus
* AF due to reversible cause
* Patients with left atrial size > 55mm or significant mitral valve disease (moderate or severe mitral stenosis or regurgitation)
* Pregnancy
* Asthma, history of bronchospasm or known adverse reaction to adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2009-12; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to first recurrence of electrocardiographically documented, symptomatic AF or atrial flutter/tachycardia between 3 and 12 months post ablation in the absence of antiarrhythmic drug therapy. | Between 3 and 12 months post ablation
  The primary outcome is time to first recurrence of symptomatic ECG-documented AF or atrial flutter/tachycardia between days 91 & 365 after ablation, or repeat ablation procedure during the first 90 days. AF or atrial flutter/tachycardia will qualify as an arrhythmia recurrence after ablation if it lasts 30 seconds or longer and is documented by 12-lead ECG, surface ECG rhythm strips, or TTM recordings. Documented episodes will be adjudicated by a blinded committee. Time 0 is defined as day 91 post ablation with FUp's extending 365 days post ablation.

SECONDARY OUTCOMES:
Time to first recurrence of any electrocardiographically documented AF or atrial flutter/tachycardia (symptomatic or asymptomatic) between days 91 and 365 after ablation. | between 3 and 12 months
Repeat ablation procedure for documented recurrence of symptomatic AF or atrial flutter/tachycardia. | between 3 and 12 months
Emergency visits or hospitalizations | between 0 and 12 months
Antiarrhythmic drug use because of documented recurrence of symptomatic AF or atrial flutter/tachycardia | between 0 and 12 months
Proportion of patients with AF or left atrial flutter/tachycardia occurring during the first 90 days post ablation | between 0 and 3 months
Major peri-procedural complications including stroke, PV stenosis, cardiac perforation, atrio-esophageal fistulae, and death | between 0 and 12 months
Generic and disease specific quality of life (assessed by the Cardiovascular Society Severity in AF (CCS-SAF) scale and SF-36 questionnaire at baseline, and at 3, 6 and 12 months post randomization). | between 0 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Macle, MD, Principal Investigator — Montreal Heart Institute
Locations (18):
- Royal Perth Hospital, Perth, Western Australia, Australia
- KH d. Elisabethinen Linz GmbH, Linz, Linz, Austria
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium
- Canada (11):
  - Foothills Medical Center, Calgary, Alberta
  - Royal Jubilee Hospital, Vancouver, British Columbia
  - QE II Health Sciences Center, Halifax, Nova Scotia
  - McMaster University and Hamilton Health Sciences, Hamilton, Ontario
  - London Health Science Centers, London, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
- Hôpital Cardiologique du Haut-Lévêque, Bordeaux, Bordeaux, France
- Germany (3):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen, Bad Krozingen
  - University Heart Center, Hamburg, Eppendorf
  - Deutsches Herzzentrum Muenchen, Munich, Muenchen

REFERENCES:
- [Derived] Willems S, Khairy P, Andrade JG, Hoffmann BA, Levesque S, Verma A, Weerasooriya R, Novak P, Arentz T, Deisenhofer I, Rostock T, Steven D, Rivard L, Guerra PG, Dyrda K, Mondesert B, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S, Macle L; ADVICE Trial Investigators*. Redefining the Blanking Period After Catheter Ablation for Paroxysmal Atrial Fibrillation: Insights From the ADVICE (Adenosine Following Pulmonary Vein Isolation to Target Dormant Conduction Elimination) Trial. Circ Arrhythm Electrophysiol. 2016 Aug;9(8):e003909. doi: 10.1161/CIRCEP.115.003909. PMID 27516462
- [Derived] Macle L, Khairy P, Weerasooriya R, Novak P, Verma A, Willems S, Arentz T, Deisenhofer I, Veenhuyzen G, Scavee C, Jais P, Puererfellner H, Levesque S, Andrade JG, Rivard L, Guerra PG, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S; ADVICE trial investigators. Adenosine-guided pulmonary vein isolation for the treatment of paroxysmal atrial fibrillation: an international, multicentre, randomised superiority trial. Lancet. 2015 Aug 15;386(9994):672-9. doi: 10.1016/S0140-6736(15)60026-5. Epub 2015 Jul 23. PMID 26211828
- [Derived] Andrade JG, Pollak SJ, Monir G, Khairy P, Dubuc M, Roy D, Talajic M, Deyell M, Rivard L, Thibault B, Guerra PG, Nattel S, Macle L. Pulmonary vein isolation using a pace-capture-guided versus an adenosine-guided approach: effect on dormant conduction and long-term freedom from recurrent atrial fibrillation--a prospective study. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1103-8. doi: 10.1161/CIRCEP.113.000454. Epub 2013 Oct 4. PMID 24097372
- [Derived] Macle L, Khairy P, Verma A, Weerasooriya R, Willems S, Arentz T, Novak P, Veenhuyzen G, Scavee C, Skanes A, Puererfellner H, Jais P, Khaykin Y, Rivard L, Guerra PG, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S; ADVICE Study Investigators. Adenosine following pulmonary vein isolation to target dormant conduction elimination (ADVICE): methods and rationale. Can J Cardiol. 2012 Mar-Apr;28(2):184-90. doi: 10.1016/j.cjca.2011.10.008. Epub 2012 Jan 2. PMID 22217936